CLINICAL TRIAL: NCT01092988
Title: A Clinical Study to Evaluate Safety of the ExAblate 2100 UF V2 System in the Treatment of Symptomatic Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Clinical Project Manager, Insightec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF032
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Uterine Fibroids; Bleeding; Pain
Keywords: Uterine Fibroids; Bleeding; Pain; Quality of life; MR guided focused ultrasound
MeSH Terms: conditions — Leiomyoma; Hemorrhage; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exablate 2100 (Experimental): MR Guided Focused Ultrasound treatment
  Interventions: Device: Exablate 2100

INTERVENTIONS:
Device: Exablate 2100 — MR guided focused ultrasound

SUMMARY:
The first magnetic resonance-guided focused ultrasound (MRgFUS) treatment of uterine fibroid using the ExAblate 2000 system was performed in 2001. Since then, more than 5000 treatments were done in more than 60 different hospitals around the world. The experience accumulated in this novel treatment was collected by InSightec and implemented into software and hardware updates, clinical tips and guidelines, all aimed to improve the clinical results and their durability, while maintaining a high level of safety.

Based on extensive clinical experience and our internal research and development effort goals toward continuous improvement in ExAblate treatment safety and performance, limited changes have been made to the current ExAblate system. This modified ExAblate system version is designated as the ExAblate 2100 UF V2 system.

The modifications are believed to improve system's friendliness to the user, without introducing new risks or other issues of safety of the device, and should not have any negative impact on the safety or technical efficacy of the treatments for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18 or older
2. Symptomatic uterine fibroids, defined as those resulting in scores of 21 or higher, based on patient responses to questions 1-8 of the Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL).
3. Women who have given written informed consent
4. Women who are able and willing to attend all study visits
5. Patient is pre or peri-menopausal (within 12 months of last menstrual period)
6. Able to communicate sensations during the ExAblate procedure.
7. Uterine fibroids, which are device accessible
8. Fibroid(s) clearly visible on non-contrast MRI.
9. Fibroid(s) enhances on MR contrast imaging

Exclusion Criteria:

1. Women who are pregnant, as confirmed by serum/urine test at time of screening, or urine pregnancy test on the day of treatment
2. Uterine size > 24 weeks
3. Patients who are breast-feeding
4. Patients with active pelvic inflammatory disease (PID).
5. Patients with active local or systemic infection
6. Contraindication for MRI Scan:

   1. Severe claustrophobia that would prevent completion of procedure in the MR unit
   2. Weight greater than 250 IBS (113Kg)
   3. Implanted ferromagnetic materials and/or devices contraindicated for MR scan
   4. Known intolerance to MRI contrast agent (e.g. Gadolinium or Magnevist)
   5. Any other contraindication for MRI Scan
7. Extensive abdominal scarring in the beam path
8. Dermoid cyst obstructing the treatment path.
9. Known pelvic malignant or pre-malignant conditions
10. Intrauterine device (IUD) anywhere in the treatment path

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety | 1 month
  Safety of ExAblate 2100 UF V2 will be determined by an evaluation of the incidence and severity of device- and procedure-related adverse events from the first visit through 1-month post-treatment.

SECONDARY OUTCOMES:
Initial Efficacy | 1 month
  Efficacy will be evaluated by comparing the Non-perfused volume obtained from this study with that of the dataset supporting PMA approval using descriptive statistics

CONTACTS AND LOCATIONS:
Locations (4):
- Radiopharmaceutiques hopital Bretonneau, Tours, France
- Sheba MC, Ramat Gan, Israel
- Research Centre of Obstetric / Gynaecology & Perinatology, Moscow, Russia
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor's website — http://www.Insightec.com